CLINICAL TRIAL: NCT06249828
Title: A Clinical Trial to Evaluate the Efficacy and Safety of Cartilage Regeneration in the Use of MegaCarti^® in Patients With Knee Joint Cartilage Injury: Multicenter, Independent Evaluator-subject Blinded, Microfracture-comparative, Randomized Clinical Study
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of MegaCarti^® in Knee Cartilage Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L&C Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LNC-MECA-004
Record Dates: First submitted 2024-01-25; First posted 2024-02-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Cartilage Defects; Microfracture; HTO; High Tibia Osteotomy; MegaCarti; Cartilage regeneration
MeSH Terms: conditions — Osteoarthritis, Knee; Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MegaCarti^® application after Microfracture Surgery (Experimental): The study group is applied with MegaCarti^® after microfracture. Afterwards, they visit at 12 weeks, 24 weeks, and 48 weeks to conduct examinations and assess Questionnaires.
  Interventions: Device: MegaCarti^®; Procedure: Microfracture
- Microfracture Surgery without Medical Devices (Active Comparator): The control group undergoes microfracture and they visit at 12 weeks, 24 weeks, and 48 weeks after surgery to conduct examinations and assess Questionnaires.
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Device: MegaCarti^® — MegaCarti® application after microfracture through athroscopic or incision surgery
  Arms: MegaCarti^® application after Microfracture Surgery
Procedure: Microfracture — Microfracture through athroscopic or incision surgery

SUMMARY:
Subjects aged 50 to 65 years with knee cartilage defects will undergo microfracture treatment for cartilage regeneration and MegaCarti^® will be applied.

DETAILED DESCRIPTION:
The MegaCarti^® is the decellularized allogeneic cartilage and acts as a cover after bone marrow stimulation to prevent the loss of blood clots and induces cartilage regeneration by assisting in the location of stem cells derived from bone marrow.

To evaluate cartilage regeneration, the study group is compared with the microfracture group alone through MOCART evaluation at 48 weeks after treatment for cartilage regeneration. In addition, a biopsy is performed to evaluate the formation of hyaline cartilage and the area ratio of regenerated cartilage is measured.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years to 65 yaers
2. After receiving a detailed explanation of this clinical trial and fully understanding it, the subject or legal representative voluntarily decides to participate in the clinical trial and sign the consent form
3. Subjects with localized full-thickness cartilage defects in the knee joint, International Cartilage Repair Society(ICRS) Grade III or IV
4. Subjects whose primary lesion site can be designated as one section of the knee joint, and the area can be determined as the main cause of clinical symptoms
5. knee cartilage defect size :1.5cm^2 to 10cm^2

Exclusion Criteria:

1. Patients who have autoimmune diseases (Ex. Rheumatoid arthritis)
2. When screening, Patients who underwent surgery related to cartilage defect treatment, such as microfracture, autologous chondrocyte therapy within the past 1 year (However, arthroscopy for diagnostic purposes is possible. Additionally, it is possible if hightibial osteotomy (HTO) has been performed in advance or is scheduled)
3. When screening, Patients who received intra-articular hyaluronic acid or steroid injections in the knee within 1 month
4. When screening, Patients who took oral steroid within 2 weeks
5. Patients who can't take MRI scan
6. BMI index : 30kg/m^2 or over
7. Patients who have gout or gout history in the knee
8. Women who are pregnant or breast-feeding, or women who have a possibility of pregnancy but do not use medically accepted methods of contraception.
9. Patients with risk factor for bleeding
10. Other than above, patients who are judged by medical investigator to be considered unsuitable for this clinical trial

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-12-13 (Actual); Study Completion 2025-12-13 (Actual)

PRIMARY OUTCOMES:
MOCART score | From 48 weeks after surgery
  The independent evaluator measure the MOCART score based on the MRI images taken at 48 weeks after surgery.
  The MOCART score is an index for evaluating the degree of restoration of cartilage tissue and consists of a total of 9 items. Each item is scored from 0 to a maximum of 20 points and added up.
  The MOCART score is 0 when the cartilage is in the worst condition, and 100 when it is in the best condition. In other words, when the clinical effect of tissue repair appears, it is evaluated as a score greater than 0.

SECONDARY OUTCOMES:
IKDC score | Baseline and 12, 24, 48 weeks after surgery
  Subjects underwent a self-assessment of knee function using the International Knee Documentation Committee Assessment (IKDC). The outcome was presented with the post-operative change amount from the baseline.
VAS | Baseline and 12, 24, 48 weeks after surgery
  Subjects underwent a self-assessment of knee joint pain using the 100-mm Visual Analogue Scale (VAS). Use of NSAIDs and acetaminophen have to be discontinued for 24 hours, respectively, prior to the VAS evaluation. The outcome was presented with the post-operative change amount from the baseline.
KOOS | Baseline and 12, 24, 48 weeks after surgery
  Subjects underwent a self-assessment of knee joint pain using the Knee Injury and Osteoarthritis Outcome score (KOOS) survey. The outcome was presented with the post-operative change amount from the baseline.
ICRS-CRA score | From 48 weeks after surgery
  Investigator uses the International Cartilage Repair Society (ICRS) - cartilage repair assessment grading (CRA) system to evaluate the degree of cartilage regeneration.
OAS | From 48 weeks after surgery
  Investigator uses the Oswestry Arthroscopic Score (OAS) system to evaluate the degree of cartilage regeneration.
Cartilage Coverage Ratio | From 48 weeks after surgery
  Using arthroscopy, the investigator calculates the area of repaired cartilage that is greater than 75% defect depth.
Histological Evaluation | From 48 weeks after surgery
  Cartilage tissue is collected from the center of the repaired knee cartilage using a needle punch. After the collected tissue is stained, an independent evaluator evaluates it using the ICRS-II Parameters evaluation sheet.

CONTACTS AND LOCATIONS:
Overall Officials: Sunghwan kim, Study Director — Yonsei University College of Medicine, Severance Hospital
Locations (7):
- South Korea (7):
  - Yonsei Sarang Hospital, Seoul, Seoul
  - Chung-Ang University Gwangmyeong Hospital, Gyeonggi-do
  - Ajou University Medical Center, Gyeonggi-do
  - Catholic Kwandong University International St.Mary's Hospital, Incheon
  - Konkuk University Medical Center, Seoul
  - Yonsei University College of Medicine, Gangnam Severance Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No